CLINICAL TRIAL: NCT03965988
Title: Effect of Docosahexaenoic Acid on Breath Holding Spells in Children: A Randomized Controlled Trial
Brief Title: Docosahexaenoic Acid on Breath Holding Spells in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: breah holding
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Breath Holding Attack
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docosahexaenoic Acid (Experimental): Docosahexaenoic acid
  Interventions: Drug: DHA
- Placebo drug (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DHA — Docosahexaenoic acid
  Other Names: Docosahexaenoic acid
  Arms: Docosahexaenoic Acid
Drug: Placebo — Placebo
  Other Names: Placebo oral tablet
  Arms: Placebo drug

SUMMARY:
DHA on Breath Holding Spells

DETAILED DESCRIPTION:
Effect of DHA on Breath Holding Spells

ELIGIBILITY:
Inclusion Criteria:

* Children with newly diagnosed sprlls

Exclusion Criteria Other treatment as iron and piracetam

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of the spells | 6 months
  Number of attacks

CONTACTS AND LOCATIONS:
Overall Officials: Amira Darwish, Lecturer, Principal Investigator — Tanta University - Faculty of Medicine; Abeer Salamah, MD, Study Director — Tanta University - Faculty of Medicine
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salamah A, Darwish AH. Docosahexaenoic Acid Plus Piracetam Versus Piracetam Alone for Treatment of Breath-Holding Spells in Children: A Randomized Clinical Trial. Pediatr Neurol. 2023 Nov;148:32-36. doi: 10.1016/j.pediatrneurol.2023.08.003. Epub 2023 Aug 9. PMID 37651975